CLINICAL TRIAL: NCT00329147
Title: A Randomized, Open-Label, Cross-Over Drug Interaction Study to Evaluate the Effects of Desvenlafaxine (DVS SR) and Paroxetine on the Pharmacokinetics of Desipramine in Healthy Subjects
Brief Title: Study Evaluating the Effects of DVS SR and Paroxetine on the Pharmacokinetics of Desipramine in Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3151A1-900
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Depression
Keywords: Healthy Subjects; Major Depressive Disorder; Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Desipramine; Paroxetine

INTERVENTIONS:
Drug: desvenlafaxine SR
Drug: desipramine
Drug: paroxetine

SUMMARY:
The purpose of this study is to evaluate the effects of multiple doses of DVS SR and paroxetine on the pharmacokinetics of a single dose of desipramine in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 18 to 55 years of age
* Healthy as determined by the investigator on the basis of medical history and physical examination, laboratory test results, vital signs, and 12-lead electrocardiogram (ECG)
* History of being a nonsmoker for at least 1 year Other inclusions apply.

Exclusion Criteria:

* Presence or history of any disorder or significant cardiovascular, hepatic, renal, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, or neurologic condition, and any severe conditions of the ears, eyes or throat (such as glaucoma or increased intraocular pressure) or psychiatric disease
* Known or suspected alcohol abuse or consumption of more than 2 standard units per day within the past 6 months
* Use of any over-the-counter, prescription, hormonal therapy or investigational medications within 30 days of study day-1 until the end of the study Other exclusions apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is to evaluate the effects of multiple doses of DVS SR and paroxetine on the pharmacokinetics of a single dose of desipramine in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Neptune City, New Jersey, United States